CLINICAL TRIAL: NCT06322849
Title: Factorial Trial Designed to Identify Active Elements of a Self-administered Digital Single-session Intervention Targeting Depressive Symptoms.
Brief Title: Active Elements of Digital Single-session Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Associate Professor, Northwestern University, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STU00220591
Record Dates: First submitted 2024-03-10; First posted 2024-03-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: Active elements; Factorial trial; Single-session interventions; Depression
MeSH Terms: conditions — Depression | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of 8 different conditions (factorial trial), following the Multiphase optimization Strategy (MOST)
Who Masked: Participant
Masking Description: Participants will be aware that they will be assigned to an intervention designed to help them with depressive symptoms. Participants will be aware that there are other arms of the study to which other participants are randomized, but they will not be aware of what these other arms entail. Additionally, the measures will be self-administered, so there is no scope for evaluator bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1 (Experimental): Experimental: Breathing exercise + active elements 1, 2, 3
  In this arm, all three factors are set to active (i.e. yes):
  * Psychoeducation
  * Testimonials and Saying is believing exercises
  * Action planning
  Interventions: Behavioral: Psychoeducation; Behavioral: Testimonials and Saying is believing exercises; Behavioral: Action planning; Behavioral: Breathing exercise
- Arm 2 (Experimental): Experimental: Breathing exercise + active elements 1, 2
  In this arm, two factors are set to active (i.e. yes):
  * Psychoeducation
  * Testimonials and Saying is believing exercises
  Interventions: Behavioral: Psychoeducation; Behavioral: Testimonials and Saying is believing exercises; Behavioral: Breathing exercise
- Arm 3 (Experimental): Experimental: Breathing exercise + active elements 1, 3
  In this arm, two factors are set to active (i.e. yes):
  * Psychoeducation
  * Action planning
  Interventions: Behavioral: Psychoeducation; Behavioral: Action planning; Behavioral: Breathing exercise
- Arm 4 (Experimental): Experimental: Breathing exercise + active elements 2, 3
  In this arm, two factors are set to active (i.e. yes):
  * Testimonials and Saying is believing exercises
  * Action planning
  Interventions: Behavioral: Testimonials and Saying is believing exercises; Behavioral: Breathing exercise
- Arm 5 (Experimental): Experimental: Breathing exercise + active element 1
  In this arm, one factor is set to active (i.e. yes):
  • Psychoeducation
  Interventions: Behavioral: Psychoeducation; Behavioral: Breathing exercise
- Arm 6 (Experimental): Experimental: Breathing exercise + active element 2
  In this arm, one factor is set to active (i.e. yes):
  • Testimonials and Saying is believing exercises
  Interventions: Behavioral: Testimonials and Saying is believing exercises; Behavioral: Breathing exercise
- Arm 7 (Experimental): Experimental: Breathing exercise + active element 3
  In this arm, one factor is set to active (i.e. yes):
  • Action planning
  Interventions: Behavioral: Action planning; Behavioral: Breathing exercise
- Arm 8 (Experimental): Experimental: Breathing exercise only
  In this arm, none of the three factors are set to active (i.e. yes)
  Interventions: Behavioral: Breathing exercise

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation is a potential active element of Project ABC. In psychoeducation, participants learn about the cognitive model of behavior and how they can take action to change their moods.
  Arms: Arm 1; Arm 2; Arm 3; Arm 5
Behavioral: Testimonials and Saying is believing exercises — Testimonials and Saying is believing exercises is a potential active element of Project ABC. In this element, participants learn about how others have taken action to improve their mood and complete one exercise where they give advice to a virtual peer who is stuck in a negative spiral.
  Arms: Arm 1; Arm 2; Arm 4; Arm 6
Behavioral: Action planning — Action planning is a potential active element of Project ABC. In this element, participants plan in detail an action they can take to get out of the negative mood spiral.
  Arms: Arm 1; Arm 3; Arm 7
Behavioral: Breathing exercise — Participants will be presented with a one-minute breathing exercise.

SUMMARY:
Depression is a leading cause of disability in young adults. However, access to care is limited due to structural and psychological barriers. Single-session interventions (SSIs) are structured programs designed to maximize the therapeutic output in one interaction between the patient and the provider or a program. Project ABC, a single-session intervention (SSI), has been shown to be effective in reducing depressive symptoms. Project ABC is based on four components-psychoeducation, testimonials, saying is believing exercises, and action planning. However, it is unclear what are the effects of the individual components.

The primary aim of this study is to calculate the main effects of the candidate components-psychoeducation, testimonials + saying is believing exercises, and action planning-on Patient Health Questionnaire-8 (PHQ-8) scores at 8-week follow-up.

The secondary aims of this study are to:

1. calculate the main effects of the candidate components-psychoeducation, testimonials + saying is believing exercises, and action planning-on PHQ-8 scores at immediate post-treatment and 2-week follow-up.
2. calculate the interaction effects, if any, among the candidate components on PHQ-8 scores at immediate post-treatment, 2-week, and 8-week follow-up.
3. calculate the main and interaction effects of the candidate components on measures of hopelessness, autonomy, relatedness, and competence.
4. determine if the effects of the candidate components on PHQ-8 are mediated by measures of autonomy, relatedness, and competence.

Additionally, the exploratory aim of this study is to determine if common factors, like credibility of the intervention and expectations to improve, can lead to symptom change.

ELIGIBILITY:
Inclusion Criteria:

* Located in the United States
* Baseline Patient Health Questionnaire-8 (PHQ-8) score >= 10
* Able to read and write English
* Able to access to the internet via a computer, tablet or smartphone for the next eight weeks

Exclusion Criteria:

* Participants who have participated in another related study on depression from our laboratory via the same participant recruitment platform in the past two months
* Participants who have submitted gibberish in open response questions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 887 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 | Baseline to 8-week post-intervention
  Patient Health Questionnaire-8 is a well-validated and self-administered measure to assess depression symptom severity in the general population. Participants are asked to rate how often they are bothered by 8 items (e.g., Poor appetite or overeating) on a scale of 0 (Not at all) to 3 (Nearly every day). Total score can range from 0 to 24, with higher scores indicating higher symptom severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-8 | Baseline to 2-week post-intervention
  Patient Health Questionnaire-8 is a well-validated and self-administered measure to assess depression symptom severity in the general population. Participants are asked to rate how often they are bothered by 8 items (e.g., Poor appetite or overeating) on a scale of 0 (Not at all) to 3 (Nearly every day). Total score can range from 0 to 24, with higher scores indicating higher symptom severity.
Beck Hopelessness Scale-4 | Baseline to immediate post-intervention; Baseline to 2-week post-intervention; Baseline to 8-week post-intervention
  Beck Hopelessness Scale-4 is the 4-item version of the 20-item Beck Hopelessness scale. Participants will be asked to rate 4 items assessing different aspects of hopelessness (e.g., My future seems dark to me) on a scale of 0 (Absolutely disagree) to 3 (Absolutely agree). Total score can range between 0 to 12 with higher scores indicating higher hopelessness.
Balanced measure of Psychological Needs scale | Baseline to immediate post-intervention; Baseline to 2-week post-intervention; Baseline to 8-week post-intervention
  The BMPN is used as a measure of the psychological needs of autonomy, relatedness, and competence as laid out by the Self-Determination Theory. It is an 18-item questionnaire where each item is rated on a scale of 1 (Strongly disagree) to 5 (Strongly agree). Scores corresponding to each psychological need will be calculated based on the items corresponding to that need. A higher score on the three needs indicates higher wellbeing. In this study, we will use a 6-item version of the scale.

OTHER OUTCOMES:
Credibility/Expectancy questionnaire | Baseline and immediate post-intervention; The second question will also be asked at 2-week post-intervention
  Two questions from Credibility/Expectancy questionnaire will be used: "At this point, how successful do you think this treatment will be in reducing your feelings of depression?" and "Over the next few weeks, how much improvement in your feelings of depression do you think will occur?" Participants will be asked to answer the questions on a scale of 1 (Not at all) to 9 (Very much).
Intervention satisfaction star rating at post-intervention | Immediate post-intervention
  Participants will be asked to rate the intervention they completed using a star rating from 1 to 5 stars, with 1 star indicating very low satisfaction and 5 stars indicating very high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available once all the planned analyses have been completed by the investigators.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and code will be made available here (https://osf.io/xbpsj/) upon publication of trial results.
Access Criteria: Will be decided on a case-by-case basis
URL: https://osf.io/xbpsj/

REFERENCES:
- [Background] Schleider JL, Mullarkey MC, Fox KR, Dobias ML, Shroff A, Hart EA, Roulston CA. A randomized trial of online single-session interventions for adolescent depression during COVID-19. Nat Hum Behav. 2022 Feb;6(2):258-268. doi: 10.1038/s41562-021-01235-0. Epub 2021 Dec 9. PMID 34887544
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Perczel Forintos D, Rozsa S, Pilling J, Kopp M. Proposal for a short version of the Beck Hopelessness Scale based on a national representative survey in Hungary. Community Ment Health J. 2013 Dec;49(6):822-30. doi: 10.1007/s10597-013-9619-1. Epub 2013 Jun 12. PMID 23756722
- [Background] Sheldon, K.M., Hilpert, J.C. The balanced measure of psychological needs (BMPN) scale: An alternative domain general measure of need satisfaction. Motiv Emot 36, 439-451 (2012). https://doi.org/10.1007/s11031-012-9279-4
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT06322849/SAP_000.pdf